CLINICAL TRIAL: NCT00384072
Title: A Multicenter, Double Blind, Randomized, Placebo Controlled Study to Assess the Safety and Efficacy of Bazedoxifene in Postmenopausal Asian Women
Brief Title: Study Evaluating the Safety and Efficacy of Bazedoxifene in Postmenopausal Asian Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3068A1-303
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-05

CONDITIONS: Postmenopause; Osteoporosis
Keywords: postmenopausal; women; SERM; osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: bazedoxifene BZA-20

SUMMARY:
The purpose of this study is to evaluate the effect of 20 mg of bazedoxifene in comparison to placebo on bone mineral density after 6 months of therapy in a population of postmenopausal Asian women.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy Asian women 45 years of age or older who are at least 1 year postmenopausal
2. Subjects must qualify for one of the following categories (a or b):

   1. Greater than 1 year but less than 5 years postmenopausal with at least one of the ospeoporosis risk factors
   2. Equal or greater than 5 years postmenopausal with BMD T-score at lumbar spine or femoral neck between -1 and -2.5 (values of -1 and -2.5 are acceptable) with at least one osteoporosis risk factor

Exclusion Criteria:

1. One (1) or more osteoporotic vertebral fractures (T4 - L4)
2. BMD T-score at the lumbar spine or femoral neck less than -2.5
3. Past history or active nontraumatic venous thromboembolic events, including deep vein thrombosis, pulmonary embolism, and retinal vein thrombosis

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The percent change from baseline in lumbar spine bone mineral density (BMD) after 6 months of treatment

SECONDARY OUTCOMES:
Additional BMD evaluation including total hip, femoral neck and trochanter at 6 months
Serum bone markers at 3 and 6 months
Lipid profile at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com
Locations (11):
- China (4):
  - Beijing
  - Nanjing
  - Shanghai
  - Tianjin
- South Korea (2):
  - Seoul
  - Suwon
- Taiwan (5):
  - Kaohsuing
  - Kaoshsuing
  - Tainan
  - Taipei
  - Tapei